CLINICAL TRIAL: NCT06695520
Title: Is the Perfusion Index an Indicator for Success of Caudal Epidural Anasthesia in Pediatric Patients?
Brief Title: Perfusion Index in Caudal Epidural Anasthesia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Monika Samir Melad, resident doctor at Anathesia , ICU & Pain Management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Perfusion Index
Record Dates: First submitted 2024-11-17; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Caudal Epidural Block
Keywords: Perfusion Index

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group (A) (Experimental): patients will receive General Anesthesia and Caudal Epidural Anesthesia
  Interventions: Procedure: Caudal epidural block
- GROUP (B) (No Intervention): patients will receive General Anesthesia only

INTERVENTIONS:
Procedure: Caudal epidural block — Ultrasound Guidance: Using ultrasound improves the accuracy of the block by allowing real-time visualization of the anatomy and needle placement . injection: .5-1mg/kg of 25% bupivacaine according to the needed block level.
  Arms: Group (A)

SUMMARY:
A caudal epidural block is among the most widely administered techniques of regional anesthesia in pediatric patients. It helps in reducing the intraoperative dose of inhalational anesthetic agent used for maintenance of anesthesia and in addition provides an excellent postoperative analgesia without the side effects of intravenous opioid medication, like nausea and vomiting during emergence, cardiovascular, and respiratory depression. the aim of the study was to assess, perfusion index (PI) as an indicator for success of caudal block onset in pediatric patients scheduled for elective surgery of lower abdomen, pelvic region, genital region, or lower limbs.

with guidance of ultrasonography.

DETAILED DESCRIPTION:
It is performed by inserting a needle through the sacral hiatus to gain entrance into the sacral epidural space. Using conventional blind technique, the failure rate of caudal epidural block is high even in experienced hands. With the advent of ultrasound in guiding needle placement, the success rate of caudal epidural block has been markedly improved and could be effective in preventing complications during caudal epidural injection. After administration of a caudal block, reliable assessment of caudal block is very crucial to ascertain the success of block. The onset of caudal block is often assessed by cold stimuli and cutaneous temperature changes. Caudal block in pediatric patients is often performed under general anesthesia. Hence, testing the sensory levels by above techniques cannot be used. Also the change in the hemodynamic parameters are few other assessment methods. These methods are to be used 15-20 min after block administration, to confirm the efficacy of a caudal block. Perfusion index (PI), independent of parameters like heart rate, oxygen saturation of blood, or body temperature, measures the ratio of arterial blood flow (pulsatile flow) to venous, capillary, and tissue blood flow (non-pulsatile blood flow) and it is shown in percentage or absolute value . PI is considered as a sensitive marker to assess the efficacy of caudal block. It can detect the onset of caudal block, by increasing PI beyond the pre-induction values, which can be due to the sympathectomy induced after successful caudal administration,which increases the blood flow to the peripheral tissues.

ELIGIBILITY:
Inclusion Criteria:

* -ASA physical status I-II. -Both sexes -Age between 2 and 10 years -Patients scheduled for elective surgery of lower abdomen, pelvic region, genital region, or lower limbs.

Exclusion Criteria:

* ASA physical status more than II.
* Patients having any neurological disorders, bleeding disorder, bony deformity of vertebral column.

infection at the injection site, drug allergy, and undergoing anal surgery.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
changes in perfusion index. | baseline
  measures the ratio of arterial blood flow (pulsatile flow) to venous, capillary, and tissue blood flow (non-pulsatile blood flow) and it is shown in percentage or absolute value

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Buono RD, Pascarella G, Costa F, Agro FE. The perfusion index could early predict a nerve block success: A preliminary report. Saudi J Anaesth. 2020 Oct-Dec;14(4):442-445. doi: 10.4103/sja.SJA_171_20. Epub 2020 Sep 24. PMID 33447184
- [Background] Kao SC, Lin CS. Caudal Epidural Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:9217145. doi: 10.1155/2017/9217145. Epub 2017 Feb 26. PMID 28337460
- [Background] Dave NM, Garasia M. A comparison of the effectiveness of predictors of caudal block in children-swoosh test, anal sphincter tone, and heart rate response. J Anaesthesiol Clin Pharmacol. 2012 Jan;28(1):17-20. doi: 10.4103/0970-9185.92428. PMID 22345939
- [Background] Xu Z, Zhang J, Shen H, Zheng J. Assessment of pulse oximeter perfusion index in pediatric caudal block under basal ketamine anesthesia. ScientificWorldJournal. 2013 Sep 19;2013:183493. doi: 10.1155/2013/183493. eCollection 2013. PMID 24174910